CLINICAL TRIAL: NCT04166617
Title: Assessment Effectiveness of the Leap Motion Capture® System on the Functionality of the Upper Limb in Acquired Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Full proffesor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01/06/2018
Record Dates: First submitted 2019-11-11; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Stroke; Treatment Adherence; Patient Satisfaction; Brain Injuries, Traumatic
MeSH Terms: conditions — Stroke; Treatment Adherence and Compliance; Patient Satisfaction; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (Active Comparator): Conventional physical therapy for upper limb in stroke patients
  Interventions: Other: Conventional therapy
- Leap motion plus conventional therapy (Experimental): Leap motion plus conventional physical therapy for upper limb in stroke patients
  Interventions: Other: Leap motion plus conventional therapya

INTERVENTIONS:
Other: Conventional therapy — conventional physcial therapy rehabilitation for the upper limb
  Arms: Conventional therapy
Other: Leap motion plus conventional therapya — leap motion plus conventional physcial therapy rehabilitation for the upper limb
  Arms: Leap motion plus conventional therapy

SUMMARY:
The affectedness of the motor control of the upper limb, particulary, the hand and/or fingers, appears in many neurological diseases, what is going to impact on the functionality of the subject. The use of new technologies in the rehabilitation environment, has the target to reduce the impact on the disabling conditions. So that, the goal of this investigation is to evaluate the system use effectiveness of the Leap Motion Controller® in the treatment on the upper limb on patients with neurological disease.

ELIGIBILITY:
Inclusion Criteria:

* people aged between 30 and 70 years old;
* with a confirmed diagnosis of brain damage (>6 months);
* UL motor impairment with a Fugl-Meyer score≥16;
* a modified Ashworth scale score≤2 in the deltoid, triceps brachii, biceps brachii and in the wrist and finger flexor and extensor muscles of the upper limb

Exclusion Criteria:

* the inability to understand instructions and actively cooperate in the tasks indicated based on a score ≥ 24 in the Mini-mental Test;
* refusal to participate in the study;
* visual impairment not correctable by glasses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-11-11 (Estimated); Study Completion 2021-11-11 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | 8 weeks
  Shoulder Pain - Physioplus Objective The Action Research Arm Test (ARAT) is a 19 item observational measure used by physical therapists and other health care professionals to assess upper extremity performance (coordination, dexterity and functioning)
Jamar | 8 weeks
  Jamar® hydraulic hand dynamometer was used to measure grip strength.
Box and blocks | 8 weeks
  Box and Blocks Test (BBT) was performed to measure unilateral gross manual dexterity in both the less and more affected side.

SECONDARY OUTCOMES:
Adherence to the therapy sessions | 8 weeks
  the attendance rate (%) for therapy sessions
Questionary of Patient Satifaction | 8 weeks
  which evaluate the level of satisfaction regarding the care and quality of the service received and the level of fulfillment of the patient's expectations regarding the treatment administered

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

REFERENCES:
- [Derived] Aguilera-Rubio A, Alguacil-Diego IM, Mallo-Lopez A, Jardon Huete A, Ona ED, Cuesta-Gomez A. Use of low-cost virtual reality in the treatment of the upper extremity in chronic stroke: a randomized clinical trial. J Neuroeng Rehabil. 2024 Jan 22;21(1):12. doi: 10.1186/s12984-024-01303-2. PMID 38254147